CLINICAL TRIAL: NCT01573182
Title: A Phase II Clinical Trial of Vaccination of Stem Cell Donors With Zostavax to Reduce the Incidence of Herpes Zoster in Transplant Recipients - A Pilot Study
Brief Title: Herpes Zoster Vaccine for Bone Marrow Transplant Donors
Acronym: VZV-Zostavax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Principal Investigator, David Gottlieb, Professor, University of Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VADOVAR
Record Dates: First submitted 2012-03-29; First posted 2012-04-06 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Herpes Zoster
Keywords: Zostavax; Herpes Zoster; VZV vaccination; Allogeneic haemopoietic stem cell transplantation
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Donor (Experimental): VZV seropositive donors 50 years and over will receive vaccination with a live attenuated herpes zoster vaccine (Zostavax) by the intramuscular (IM) route 4 to 6 weeks prior to stem cell harvesting..
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: Zostavax — VZV seropositive donors 50 years and over will receive vaccination with a live attenuated herpes zoster vaccine (Zostavax) by the IM route 4 to 6 weeks prior to stem cell harvesting.

SUMMARY:
The purpose of this study is to determine whether vaccination of stem cell donors with Zostavax can reduce the rate of Herpes Zoster reactivations in transplant recipients.

The clinical hypotheses is: 1) that Zostavax given to stem cell donors will induce protective VZV specific T cell proliferation in allogeneic stem cell transplant recipients that can be transferred to recipients; 2) and that donor vaccination with Zostavax is safe for transplant recipients as measured by viral load measurement by polymerase chain reaction assay (PCR) at the time of stem cell donation.

DETAILED DESCRIPTION:
Infection is a major cause of morbidity and death among haemopoietic stem cell transplantation patients (HSCTs). Beyond the initial post-transplant (BMT) phase of neutropenia, the most common infections are cytomegalovirus (CMV) and fungal infections. Another common infection for which BMT patients are at increased risk is varicella-zoster virus (VZV) (both primary varicella and herpes zoster). VZV infection is controlled by specific T cell responses that are impaired post stem cell transplant.

Heat inactivated VZV vaccine has been shown to more than halve the incidence of herpes zoster in adult BMT patients undergoing autologous transplantation. Clinical protection was correlated with in vitro CD4 T-cell proliferation in response to varicella-zoster virus. Being a live vaccine, attenuated VZV and (herpes zoster (HZ) vaccines are contraindicated within 24 months after allogeneic HSCT. However, priming of donor T-cells with herpes zoster vaccine may be a feasible alternative. One possible complication is the transfer of live virus from vaccinated donors to immunocompromised stem cell transplant recipients.

Normal donors donating for HLA matched siblings will be vaccinated with the Varivax vaccine prior to donation. Stem cell products will be assessed at the time of donation for evidence of VZV by PCR and for response to vaccination by T cell proliferation. Transfer of VZV proliferative responses in transplant recipients will be assessed by VZV specific T cell proliferation at 3, 6, 9 and 12 months post transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic HSCT Recipient-donor pair
* Donor aged 50 years and over
* Recipients and donors willing to be recruited as a pair to this study
* Recipients undergoing myeloablative or non myeloablative non T cell depleted, allogeneic stem cell transplants from HLA identical or 1 HLA antigen mismatched siblings.

Exclusion Criteria:

* Lack of informed consent
* Inability to recruit donor and recipient as a pair
* Autologous transplant
* Contraindication to Zostavax in donor
* Donor aged <50 years
* Recipient VZV immunoglobulin G (IgG) negative pre-transplantation,
* Donor VZV IgG negative
* Pregnancy of donor at randomisation
* Inability to follow study protocol (donor and recipient)
* Malignancy or immunosuppression of HSC donor
* Expected HSCT within 30 to 42 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Percentage of transplant recipients with VZV specific T cell proliferation within the first 12 moths post-transplant. | incidence of VZV specific T cell proliferation in the first 12 months post allogeneic stem cell transplant in recipients receiving stem cells from Zostavax vaccinated donors
  VZV specific T cell proliferation will be assessed at 3, 6, 9 and 12 months post transplant in stem cell transplant recipients.

SECONDARY OUTCOMES:
Donor VZV positivity by PCR and genotype and donor VZV specific T cell response to vaccination | 4 to 6 weeks after vaccination
  Donor VZV positivity by PCR and VZV specific T cell proliferation will be assessed 4 to 6 weeks after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: David Gottlieb, Principal Investigator — Westmead Hospital
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia